CLINICAL TRIAL: NCT03753802
Title: Multicenter Randomized Controlled Trial: Evaluation of the Effects of Respiratory Physiotherapy, Placebo-controlled, in Infants With Moderate Acute Bronchiolitis
Brief Title: Evaluation of the Effects of Respiratory Physiotherapy in Infants With Moderate Acute Bronchiolitis
Acronym: Bronkiville
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Réseau Kinésithérapie Bronchiolite Essonne (Other)
Responsible Party: Principal Investigator, Aurore TREBUCHET, Clinical Manager, Réseau Kinésithérapie Bronchiolite Essonne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-A00946-49
Record Dates: First submitted 2018-10-29; First posted 2018-11-27 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Acute Bronchiolitis
Keywords: Bronchiolitis; Chest physiotherapy; Infants
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: The treated group will receive respiratory physiotherapy treatment using slow extended and passive expiratory maneuvers. The control group will not receive physiotherapy treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be performed by the study website and will be only known by the physiotherapist. The parents are not allowed to be in the room of physiotherapy during the physiotherapy session. They don't know which treatment is allocated to their child. The evaluator physician doesn't know which treatment is allocated to the child. The biostatistician doesn't know which treatment is allocated to which group during the analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated (Experimental): The treated group will receive chest physiotherapy treatment using slow extended and passive expiratory maneuvers.
  Interventions: Other: Chest Physiotherapy
- Control (Placebo Comparator): The control group will not receive physiotherapy treatment.
  Interventions: Other: Surveillance

INTERVENTIONS:
Other: Chest Physiotherapy — During sessions, the child is lying on the back, he should not have eaten within two hours prior to the sessions. An extended slow expiration handling is performed on 3 respiratory cycles consecutive, this session is repeated for 10 minutes. Breaks are made regularly during the treatment to have approximately 5 to 6 minutes of handling and 4-5 minutes of rest on the total 10 minutes of treatment. Induced cough handlings will be conducted at five minutes and at ten minutes if the child has not coughed during the movements of chest physiotherapy. These are performed by a brief pressure above the jugular (suprasternal) notch of the patient. Only two consecutive trials of the induced cough handling are allowed, even if the handlings are unsuccessful the physiotherapist does not insist. The following 5 minutes of the session are 5 minutes of rest. During the sessions the physiotherapist wears a mask and respects the usual rules of hygiene.
  Arms: Treated
Other: Surveillance — The session is only a surveillance session with the physiotherapist. The physiotherapist is only watching over the child. The parents of the child wait in the waiting room during the physiotherapy session. They don't know which treatment (chest physiotherapy or no treatment) is applied to their child.
  Arms: Control

SUMMARY:
Bronchiolitis affects 460,000 children in France per year. The French study called "Bronkilib 2" found a positive effect of chest physiotherapy treatment. This study and the work done so far in chest physiotherapy prompt us to recommend respiratory physiotherapy with slow passive expiratory handlings in the treatment of the moderate bronchiolitis of infants. But, further studies are still needed to corroborate these early findings. The Cochrane is recommending new high-level proof studies on passive expiratory techniques to conclude about their benefits.

The aim of this study is to evaluate the effectiveness of the bronchial drainage procedure carried out during chest physiotherapy sessions, during episodes of moderate to acute bronchiolitis in infants aged 3 to 24 months. Currently, the French High Authority for Health recommends performing physiotherapy sessions for the symptomatologic treatment of acute bronchiolitis in infants - in cases where it could be described as moderate - but few studies have demonstrated the efficacy of this treatment.

The study included infants with a first or a second episode of bronchiolitis classified as moderate according to the Wang's Respiratory score. The treated group will receive chest physiotherapy treatment using slow extended and passive expiratory handlings. The control group will not receive physiotherapy treatment. The study will be conducted during 4 days. The clinical symptoms and the general health condition of the infant will be evaluate by questionnaires.

DETAILED DESCRIPTION:
Bronchiolitis affects 460,000 children in France per year. The French study called "Bronkilib 2" found a positive effect of chest physiotherapy treatment. This study and the work done so far in chest physiotherapy prompt us to recommend respiratory physiotherapy with slow passive expiratory handlings in the treatment of the moderate bronchiolitis of infants. But, further studies are still needed to corroborate these early findings. The Cochrane is recommending new high-level proof studies on passive expiratory techniques to conclude about their benefits.

The aim of this study is to evaluate the effectiveness of the bronchial drainage procedure carried out during chest physiotherapy sessions, during episodes of moderate to acute bronchiolitis in infants aged 3 to 24 months. Currently, the French High Authority for Health recommends performing physiotherapy sessions for the symptomatologic treatment of acute bronchiolitis in infants - in cases where it could be described as moderate - but few studies have demonstrated the efficacy of this treatment: the only randomized trial on French techniques of chest physiotherapy concerning outpatients is "Bronkilib 2", pending publication. It is therefore the second such study in France that will corroborate or invalidate the results of the "Bronkilib 2" study.

The study included infants with a first or a second episode of bronchiolitis classified as moderate according to the Wang's Respiratory score (3 <score <9). The treated group will receive chest physiotherapy treatment using slow extended and passive expiratory handlings. The control group will not receive physiotherapy treatment. To control parents' home care and ensure comparability of groups, an education session to the rhinopharyngeal clearance procedure will be conducted in both groups.

The study will be conducted during 4 days per participant. The study will evaluate the Wang's Respiratory score change measured between day 1 and day 4 and the evolution of the general health condition of the infant between sessions. The study will also evaluate the saturation, the results of a human Respiratory Syncytial Virus (RSV) nasal swab test, and the "inflamed / secretory" status of children. The Wang's Respiratory score, the saturation and the inflamed/secretory status will be collected through questionnaires available on the website of the study. The general health condition of the infants will be collected by the QUALIN questionnaire given to the parents.

The study will be conducted as follow:

A study session begins on Friday of week 0, children may be included on Monday or Tuesday of the following week (week 1). The session ends on the next Friday (week 1). Children entered on Monday are seen until Thursday, children entered on Tuesday are seen until Friday. Children can have a prescription dating back to Monday or Tuesday, or the previous week (Friday or Saturday).

The day 0 is the day where the child is greeted by the prescribing physician, general practitioner or paediatrician of the family. Its role is to inform the parents of the child of the existence of the study. This includes: checking the criteria of inclusion and exclusion, including Wang's Respiratory score; explaining the course of the study; providing the patient with an information letter, a consent letter and letters of no objection; giving him the treatment prescription; giving them the access information to the center and the phone number of the physiotherapist (which they have to call without delay on the first scheduled day); and answering their questions.

Parents have the right to a cooling-off period (minimum 1 hour). Nevertheless, the entry in the study cannot occur after Tuesday of the study week, and without prior consultation with other physiotherapists. Parents wishing to integrate the study are to call the physiotherapist indicated by the prescribing physician for an appointment.

Day 1 is a Monday or a Tuesday. The child is greeted by the physiotherapist who is expected to: schedule the appointment with the parents either by phone or in person, collect at least a consent letter, collect the letters of no objection, answer the questions of parents, remind that the consent of both legal guardians is required, if not the case inform them that they will be re-contacted by the principal investigator due to this missing writing consent. Then the physiotherapist has to enter the child name in the database via the study website to receive the child code which will be given to the parent. Thus, the child gets a code which will be then the only way to recognize him/her. The physiotherapist asks the evaluating physician to evaluate the Wang's Respiratory score of the day 1.

The evaluating physician comes into the physiotherapy room to: check that the child meets the criteria for inclusion in the study (no worsening of the general condition and Wang's Respiratory score < 9), evaluate the first assessment by the Wang's Respiratory score. This evaluation is filled on the study website with the identifiers of the physician and the child. Then the physician leaves the room.

Then, the physiotherapist performs the RSV nasal swab test. He has the parents perform the rhinopharyngeal clearance to verify that the procedure is known and correct. He gives the QUALIN questionnaire to the parents. He then asks the parents to leave the room for the session and asks the website to randomize the treatment. The treatment to be applied is then displayed on the screen, it is visible on the page dedicated to physiotherapists. Physicians have no access to this information. Then the physiotherapist performs the treatment provided by the randomization.

Randomization is performed at this time in order to avoid a randomization of treatment on children who would get out of the study before the session of physiotherapy, which would create a risk of imbalance between upstream groups.

During the physiotherapy session, parents in the waiting room fill in the QUALIN questionnaire they will hand over to the physiotherapist after the session. Parents are not present in the physiotherapy room during the sessions. The physiotherapist fills balance sheets of saturation for all children and the status of the child (inflamed / secreting) for children in the treatment group.

Day 2, 3 and 4 the child is seen again by the evaluating physician for a Wang's Respiratory score: prior to the session of physiotherapy or surveillance for days 2 and 3, 30 minutes after the session for the day 4. The balance sheets of saturation (at T30 the day 4) and status of the child (inflamed / secreting) are again filled by the physiotherapist. The parents fill in the questionnaire QUALIN in the waiting room during sessions.

Day 4, the study session is over. The evaluating physician suggests the continuation or cessation of sessions of chest physiotherapy, depending on the health state of the child during its last evaluation of the Wang's Respiratory score.

Evaluating physicians and physiotherapists are present from Monday to Friday (13 h to 19 h). Each Center has at least one physician present every day during this period. Each Center has a physiotherapist on call every day during this period.

The side effects or the non presentation of the child at the session can be collected at any time of the study by: the evaluating physician and physiotherapist on the study website and via the dedicated tab. The information is then sent directly to the proponent, the principal investigator and coordinating physician. If there is a hospitalization, an emergency unblinding can be made by the proponent, the principal investigator or the Coordinating doctor who will be notified by mail and phone: the guardians are informed by mail and/or phone of the treatment received and results of the assessments made.

If the child is getting worse: if Wang's Respiratory score ≥ 9 or if the child's condition becomes cause for concern during the assessment carried out by the evaluating physician (child receptive, amorphous, signs of respiratory distress associated with a frequency respiratory > 60 breaths / minutes, signs of cyanosis, saturation ≤ 94%), the child must be taken out of the study and sent to a hospital. If this takes place during the session of physiotherapy, physiotherapist must ask the evaluating physician an assessment. An emergency unblinding is made by the proponent, the principal investigator or coordinating physician.

These criteria of aggravation are recalled on the study website when filling out the balance sheet by therapists. If the criteria are met the site visually alerts the therapist and suggests him to go to the 'side effects' tab. The physiotherapist and the evaluating physician can at any time report such signs.

If one of the guardians wishes to get out of the study, he informs the evaluating physician or the physiotherapist or some other official who report it on the study website. The reason for getting out of the study will be sought by the principal investigator without pressure. Legal guardians have the right to wish not to report the reason why they get out of the study. If the child is not present at the scheduled appointments or during the day, this will be reported by the physiotherapist since it will take the child out of the study.

It is expected to treat 168 subjects, that is to say 84 subjects per group, over the two medical centers. This will allow to perform the statistical analyses (Chi2). The number of subjects has been estimated based on the results of the French "Bronkilib 2" study and Postiaux study.

The results will be presented in descriptive statistics by diagrams and box plots. The inferential statistics used will be: the Chi2 test to evaluate the intensity of the change in the Wang's Respiratory score between day 1 and day 4, the Logrank test to evaluate the change in the general health condition of the child (QUALIN questionnaire) during the four days of the study, the Smirnov test to evaluate the change in the oxygen saturation during the four days of the study. The Chi2 test will be performed using stratification on RSV status and inflamed/secretory status. A Principal Components Analysis will be performed to identify which items of the QUALIN score (so of the general health condition of the child) have been impacted by the chest physiotherapy. The potential relation between the Wang's Respiratory score and the QUALIN questionnaire will be estimated by the Kendall correlation coefficient. Missing data will be estimated by imputation, either using prior data or information collected on why the participant got out of the study.

The study can be stopped at any moment by the French Committee for the Protection of Persons (CPP), or by the French Authority for Medication and Biomedical Research (ANSM).

ELIGIBILITY:
Inclusion Criteria:

* Acute bronchiolitis diagnosed during a medical consultation in one of the centres and medical agreement: the prescription must be based on clinical diagnosis of bronchiolitis proposed by the Guideline of the Academy of Pediatrics (AAP), i.e. the presence of rhinorrhea, cough, wheezing or rales crinkly, tachypnea, intercostal or chest indrawing, use of accessory muscles, flapping of the wings of the nose, expiratory grunting, lowest oxygen saturation (strictly less than 95%). The presence of three of these signs is enough to make the diagnosis of infant acute bronchiolitis.
* First or second episode of bronchiolitis: three episodes of bronchiolitis in the same winter suggest infant asthma, or the presence of other respiratory disease. To avoid any selection bias which might have a negative impact on the results of the study, only the first or second episode of bronchiolitis will be included.
* 3 months ≤ age ≤ 24 months: children of less than three months have a very immature lung. To avoid any worsening of the health condition of the child, related to potential but not considered side effects of the treatment, the study will be conducted on children over 3 months old.
* 3 < Wang's score < 9: bronchiolitis is considered light when Wang's score is less than or equal to 3 and as severe when Wang's score is greater than or equal to 9. The French Health Authority and the Cochrane discourage chest physiotherapy for the treatment of severe bronchiolitis. A hospital medical support is more adequate than a liberal support for this type of patient. They will not be included in the study.
* Informed written consent of the holders of parental authority: an information and consent form will be read and explained to the holders of parental authority before collecting their written consent during the interview with the prescribing physician. Consent will be collected by the physiotherapist on call of the investigative Centre, to let a cooling-off period for the holders of parental authority.

Exclusion Criteria:

* Refusal of parents or holders of parental authority.
* No medical prescription: will only be included in the study children whose health can in no respect be endangered by their inclusion.
* Comorbidities: cardiac, pulmonary, neurological disease, immunodeficiency, congenital anomaly, other diseases explaining respiratory symptoms: the presence of comorbidities is likely to introduce a selection or a confusion bias in the results of the study. These patients will not be included in the study.
* Wang's score ≤ 3 or ≥ 9: a score ≥ 9 requires a hospitalization.
* Status of the child requiring hospitalization.
* No affiliation to a social security scheme.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of the Wang's Respiratory score between day 4 and day 1 | Each day, before the physiotherapy session for the day 1 to 3, after for the day 4.
  The Wang's Respiratory score as previously described in the literature by Wang E.E, measures the clinical state of the child. It includes 4 items : respiratory rate (breaths/minute ; quoted from 0 to 3), wheezing (quoted from 0 to 3), retraction (quoted from 0 to 3) and general condition (quoted from 0 or 3). The Wang's Respiratory score quotes the clinical state of the child from 0 to 12, the clinical state being normal for a score of 0, and worrying for a score greater than or equal to 9.
Time from the date of first measure until the date of first documented improvement (up to 4 days), defined as an increase of 10 points from the QUALIN score (for child under 24 months age old) compared to the initial score. | Time from the date of first measure until the date of first documented improvement (up to 4 days), defined as an increase of 10 points from the QUALIN score (for child under 24 months age old) compared to the initial score.
  The QUALIN score measures the general health condition and the quality of life of the child. It will be fill out by the parents. The QUALIN score contains 34 items, evaluating the awakening state, the psychological and somatic behavior of the child. Each item can be quoted by the parents from completly true to completly false. The total score quotes the quality of life of the child from -68 to +68, a negative score meaning that the child have a poor general health condition and quality of life, a positive score meaning that the child have a good general health condition and quality of life.

SECONDARY OUTCOMES:
Change in Oxygen saturation between day 4 and day 1, and between day 2 and day 1 | Each day, before the physiotherapy session for the day 1 to 3, after for the day 4.
  Oxygen saturation estimate by a pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BAUCHER, Principal Investigator — Réseau Kinésithérapie Bronchiolite Essonne
Locations (3):
- France (3):
  - Maison de Santé Pluri professionnelle Les allées, Corbeil-Essonnes, Essonne
  - Cabinet Pédiatrique Saint-Germain, Saint-Germain-lès-Arpajon, Essonne
  - MSP Léonie Chaptal, Athis-Mons

IPD SHARING:
Plan to Share IPD: Yes
Collected individual participant data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: Collected individual participant data shared upon request for Meta-analyses or other publications, co-decided by the sponsor (RKBE) and the investigators of the study.

REFERENCES:
- [Background] Postiaux G, Louis J, Labasse HC, Gerroldt J, Kotik AC, Lemuhot A, Patte C. Evaluation of an alternative chest physiotherapy method in infants with respiratory syncytial virus bronchiolitis. Respir Care. 2011 Jul;56(7):989-94. doi: 10.4187/respcare.00721. Epub 2011 Feb 22. PMID 21352671
- [Background] Remondini R, Santos AZ, Castro Gd, Prado Cd, Silva Filho LV. Comparative analysis of the effects of two chest physical therapy interventions in patients with bronchiolitis during hospitalization period. Einstein (Sao Paulo). 2014 Oct-Dec;12(4):452-8. doi: 10.1590/S1679-45082014AO3230. PMID 25628196
- [Background] S Goncalves RA, Feitosa S, de Castro Selestrin C, Valenti VE, de Sousa FH, F Siqueira AA, Petenusso M, de Abreu LC. Evaluation of physiological parameters before and after respiratory physiotherapy in newborns with acute viral bronchiolitis. Int Arch Med. 2014 Jan 8;7(1):3. doi: 10.1186/1755-7682-7-3. PMID 24401198
- [Background] Postiaux G, Zwaenepoel B, Louis J. Chest physical therapy in acute viral bronchiolitis: an updated review. Respir Care. 2013 Sep;58(9):1541-5. doi: 10.4187/respcare.01890. Epub 2013 Jan 3. PMID 23287014
- [Background] Pupin MK, Riccetto AG, Ribeiro JD, Baracat EC. Comparison of the effects that two different respiratory physical therapy techniques have on cardiorespiratory parameters in infants with acute viral bronchiolitis. J Bras Pneumol. 2009 Sep;35(9):860-7. doi: 10.1590/s1806-37132009000900007. English, Portuguese. PMID 19820812
- [Background] Sanchez Bayle M, Martin Martin R, Cano Fernandez J, Martinez Sanchez G, Gomez Martin J, Yep Chullen G, Garcia Garcia MC. [Chest physiotherapy and bronchiolitis in the hospitalised infant. Double-blind clinical trial]. An Pediatr (Barc). 2012 Jul;77(1):5-11. doi: 10.1016/j.anpedi.2011.11.026. Epub 2012 Jan 26. Spanish. PMID 22281403
- [Background] Ralston SL, Lieberthal AS, Meissner HC. Ralston SL, Lieberthal AS, Meissner HC, et al. Clinical Practice Guideline: The Diagnosis, Management, and Prevention of Bronchiolitis. Pediatrics. 2014;134(5):e1474-e1502. Pediatrics. 2015 Oct;136(4):782. doi: 10.1542/peds.2015-2862. No abstract available. PMID 26430140
- [Background] Roque i Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2016 Feb 1;2(2):CD004873. doi: 10.1002/14651858.CD004873.pub5. PMID 26833493
- [Background] Wang EE, Milner RA, Navas L, Maj H. Observer agreement for respiratory signs and oximetry in infants hospitalized with lower respiratory infections. Am Rev Respir Dis. 1992 Jan;145(1):106-9. doi: 10.1164/ajrccm/145.1.106. PMID 1731571
- [Background] Gomes GR, Calvete FP, Rosito GF, Donadio MV. Rhinopharyngeal Retrograde Clearance Induces Less Respiratory Effort and Fewer Adverse Effects in Comparison With Nasopharyngeal Aspiration in Infants With Acute Viral Bronchiolitis. Respir Care. 2016 Dec;61(12):1613-1619. doi: 10.4187/respcare.04685. Epub 2016 Aug 23. PMID 27555618
- [Background] Manificat S, Dazord A, Langue J, Danjou G, Bauche P, Bovet F, Cubells J, Luchelli R, Tockert E, Conway K. [Evaluation of the quality of life of infants and very young children: validation of a questionnaire. Multicenter European study]. Arch Pediatr. 2000 Jun;7(6):605-14. doi: 10.1016/s0929-693x(00)80127-x. French. PMID 10911526
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocole, SAP and ICF (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT03753802/Prot_SAP_ICF_002.pdf